CLINICAL TRIAL: NCT01099111
Title: Advanced Metagenomic Analysis of Human Colonic Microbiota in Patients With Chronic Gastrointestinal Disorders (IBS, IBD, CRC)
Brief Title: Advanced Metagenomic Analysis of Human Colonic Microbiota in Patients With Chronic GI Disorders
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Ahmed Al Omair, Head, GI section + GI Consultant, King Fahad Medical City
Other Study IDs: 09 -116; 243 - 29 - AT (Other Grant/Funding Number: KACST (Saudi Arabia))
Record Dates: First submitted 2010-04-01; First posted 2010-04-06 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Irritable Bowel Syndrome; Colitis, Ulcerative; Crohn Disease; Colonic Neoplasms
Keywords: IBS; UC; CD; CRAP/CRC
MeSH Terms: conditions — Irritable Bowel Syndrome; Colitis, Ulcerative; Crohn Disease; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colonic washing samples from 4 specific segments (cecum, transverse, proximal sigmoid and rectum) of every subject will be retained for 16S rRNA analysis for the study purpose, and more samples will be retained for further analysis later on.
  Samples from the unified colonic segments (each collected as 15 cc in each of four 20 cc tubes and stored in -70 Freezer) were completely recruited from 50 normal subjects, 50 IBS, 50 UC, 46 CD and only 29 CRC.
  One to two tubes from each segment sample of all subjects have been utilized for DNA extraction and accepted if identified sufficient according to lab. Hence submitted for 16S rRNA analysis. Currently we are waiting for intra-cohort comparison of samples, then inter-cohort comparisons among different study groups will be done.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Irritable Bowel Syndrome: only one Colonoscopy with mucosal washing samples collection at the time of recruitment
- Ulcerative Colitis: only one Colonoscopy with mucosal washing samples collection at the time of recruitment
- Crohn's Disease: only one Colonoscopy with mucosal washing samples collection at the time of recruitment
- Colo Rectal Cancer: only one Colonoscopy with mucosal washing samples collection at the time of recruitment
- Control: Normal Subjects: only one Colonoscopy with mucosal washing samples collection at the time of recruitment

SUMMARY:
This clinical trial hypothesize that Gut Microbiota (bacteria, viruses, fungi)play a major role in the occurrence and progression of many chronic gastrointestinal diseases like Irritable Bowel Syndrome, Inflammatory Bowel Diseases and Colo-Rectal Cancer.

Hence, aims to study the spectrum of such microbiota in these patients as compared to normal subjects, by utilizing metagenomic techniques rather than cultural methods.

DETAILED DESCRIPTION:
The terms intestinal "microflora" or "microbiota" refer to the microbial ecosystem colonizing the gastrointestinal tract. Recently developed molecular biology instruments suggest that a substantial part of bacterial communities within the human gut still have to be described. Intestinal bacteria play an essential role in the development and homeostasis of the immune system. Most of these important microbiota are unculturable which significantly have limited our understanding of bacterial-host crosstalk. Among the methods designed to gain access to the physiology and genetics of uncultured organisms, metagenomics, the genomic analysis of a population of microorganisms, has emerged as a powerful technology. Metagenomics is the study of genomic content in a complex mixture of microorganisms. Direct isolation of genomic DNA from an environment circumvents culturing the organisms under study. The two primary goals of this approach are to develop a consensus of what populations of microorganisms are present and then to identify what roles each microorganism has within a specific environment. Metagenomics samples are found nearly everywhere, including several microenvironments within the human gut, soil samples, extreme environments such as deep mines and the various layers within the ocean. Therefore, the diversity of microorganisms is thought to be in the range of hundreds of millions to greater than tens of trillions of species. Among the most mysterious microenvironment is the human gastrointestinal tract that harbor greater than thousands of millions of microbial species (at least 1014), including up to 2000 species dominated by anaerobic bacteria.

Many of the gastrointestinal or even other diseases (metabolic as in obesity, or autoimmune as in allergies) involve primarily the human gut microbiota and then according to specific changes in microbiota equilibrium certain effects occur on either bowel motility (as in irritable bowel syndrome: IBS), homeostasis of the GI immune system (as in inflammatory bowel disease: IBD), or mucosal cells proliferation (as in adenoma - colorectal cancer: CRC). These chronic diseases affect all nations worldwide and represent a significant public health burden. They can be seen among children, adolescents, and adults. Currently there is no medical cure for IBS, IBD or CRC once they develop.

The complex interactions between microbial, genetic, immune, and environmental factors seem to play an important role in the pathogenesis of IBS, IBD and CRC. Lately, post infectious - IBS have gained increasing focus, to the extent that whole pathogenesis of IBS might be attributed to a specific triggering factor of microbiota imbalance. The prevailing theory is that IBD is related to an altered mucosal barrier with a deregulated immune response directed against specific modifications in the normal microbiota leading to the alteration of its equilibrium. The etiology of IBD can therefore be conceptualized as an aberrant immunologic response to a modified component or components of the gut microbiota potentially following an environmental insult. Likewise, CRC development process from normal mucosal surface to adenoma and finally to CRC; is probably related to gut microbiota.

The prevalence of these diseases has been documented to go through an obvious increase in Saudi Arabia during the last 3 decades. This would represent a unique model to study the role of GIT microbiota or their metagenomics and their modifications in response to environmental or dietary factors in this community that went into urbanization fairly recently, and then analyze their causative relations to the focus diseases.

Here, we propose to perform a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis in normal subjects and patients with IBS, IBD and CRC by using state of the art metagenomics technology. This will be done on a Saudi population sample that we believe represent a unique model.

Our specific objectives for this project are:

* Characterize the microbiota composition (microbes and virus) of the mucosa from Saudi patients with IBS, IBD and CRC.
* Characterize the mobile GI metagenomics of Saudi patients with IBS, IBD and CRC.
* Compare the metagenomics of IBS, IBD and CRC patients to each other and to normal subjects from the same population.

Expected outcomes and Significance of research:

Altogether, the results from aims 1 and 2 will provide for the first time a comprehensive and in-depth analysis of the mucosa-associated microbiota of adult patients with IBS, IBD and CRC in Saudi population. The proposed study will define a microbiota "fingerprint" for Saudi norms, IBS, IBD and CRC. The contribution of virome and the mobile metagenome into these diseases development and/or health maintenance will be assessed for the first time and thus has the potential to reveal new paradigms. In addition, the study of the virome and mobile metagenome will help us to understand the selective forces that could contribute to the alteration and evolution of the microbiota community and thus could have important implications for the treatment of the diseases. Certainly, the work proposed here will pave the way toward future hypothesis-driven research which could lead to the design of therapeutic strategies aimed at manipulating the microbial community.

ELIGIBILITY:
Inclusion Criteria:

IBS: 50 consecutive patients presenting to KFMC GI service after launching the project on July 2010, will be recruited if they meet the following conditions:

1. Meet the diagnostic criteria as per ROME-II classification and as judged by experienced consultants for not less than 5 years.
2. IBS with diarrhea or constipation or mixed predominance pattern will be included.
3. Standard diagnostic tests have to be done to exclude any possible organic lesion to explain the abdominal pain, and all have to be negative.

IBD: from the KFMC GI service database, 50 Ulcerative Colitis (UC) and 50 Crohn's Disease (CD) will be selected according to following:

1. Confirmed diagnosis as CD or UC based on clinical, endoscopic and histological criteria.
2. Specifically did not use antibiotics for last 6 months before enrollment.
3. Detailed information about current treatment regimen has to be provided, and current use of 5-ASA, Steroid or Azathioprine will not hold from enrolling the patients as we cannot have patients off any one or more of these medications. (Obviously, we cannot exclude effects of these medications on microbiota, but it is not the focus of the current study).
4. None of the patients selected would be on anti-TNF medications.

CRC: 50 consecutive cases of confirmed CRC as per histological diagnosis made by 2 experienced pathologists will be included. Feasibility to do full colonoscopy before any surgical resection would be a condition to recruit any patient.

Normal Subjects: 50 normal control groups that are matched for age and sex to the other 3 disease groups will be selected from consecutive CRC screening colonoscopy subjects who get referred to KFMC GI service during the study period, and proved to have no GI disorders. 25 will be selected from Urban and 25 from Rural areas of KSA.

Exclusion Criteria:

1. Treatment with antibiotics for the last 6 months before enrollment.
2. Absence of recent infective colitis, bowel obstruction, or colonic/small intestinal resection surgery.
3. Not on any medication that may affect gut microbiota, like: cholestyramine, ursodeoxycholic acid, gut prokinetic agents.
4. Refusal to comply with the unified bowel preparation instructions for all cases.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We propose to recruit our cohort of patients from the King Fahad Medical City in Riyadh (largest tertiary care hospital of Saudi MOH with wide open referral system), over one year between July 2010 and July of 2011. Fifty participants with each of the focus conditions (IBS, UC, CD, CRC) will be compared to fifty participants with no GI complaints and have a normal colonic mucosa (by endoscopic and histological examination).
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O AlOmair, MD, Principal Investigator — KFMC; Ali Al Shanqeeti, MD, Study Chair — KACST
Locations (1):
- KFMC, Riyadh, Riyadh Region, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at KFMC (tertiary care medical center), starting 1/7/2010 and completed 29/9/2012. Demographic and clinical data were collected for all, together with performance of colonoscopy at entry and collection of samples as specified.
Pre-assignment Details: We were able to recruit the desired number for normal, IBS and UC groups. However, in view of strict inclusion and exclusion criteria, only 46 were recruited for CD and only 29 were recruited for CRC.
  Moreover, DNA extraction was not sufficient for some subjects at all groups that indicate replacing them with other patients.
Groups:
- Irritable Bowel Syndrome: 50 subjects that exactly meet our inclusion & exclusion criteria were recruited. Demographic and clinical data were entered for each during the introduction to the study and verifying acceptance to participate. Then after unified bowel preparation protocol, a full Colonoscopy was performed after signing the consent, during which mucosal washing samples were collected from the unified 4 colonic segment sites, as specified in methodology.
  Recruitment were completed on 08/05/2011, however, in view of insufficient DNA extraction of 5 subjects they have been replaced (on 28/07/2012) with other 5 subjects following exactly the same protocol.
  Now, all are identified as sufficient DNA extraction and had been enrolled into a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis by using state of the art metagenomics technology.
- Ulcerative Colitis: 50 subjects that exactly meet our inclusion & exclusion criteria were recruited. Demographic and clinical data were entered for each during the introduction to the study and verifying acceptance to participate. Then after unified bowel preparation protocol, a full Colonoscopy was performed after signing the consent, during which mucosal washing samples were collected from the unified 4 colonic segment sites, as specified in methodology.
  Recruitment were completed on 05/06/2012, however, in view of insufficient DNA extraction of 3 subjects they have been replaced on 16/09/2012 with other 3 subjects following exactly the same protocol.
  Now, all are identified as sufficient DNA extraction and had been enrolled into a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis by using state of the art metagenomics technology.
- Crohn's Disease: 46 subjects that exactly meet our inclusion & exclusion criteria were recruited. Demographic and clinical data were entered for each during the introduction to the study and verifying acceptance to participate. Then after unified bowel preparation protocol, a full Colonoscopy was performed after signing the consent, during which mucosal washing samples were collected from the unified 4 colonic segment sites, as specified in methodology.
  Recruitment were completed on 27/05/2012, however, in view of insufficient DNA extraction of 2 subjects they have been replaced on 05/09/2012 with other 2 subjects following exactly the same protocol.
  Now, all are identified as sufficient DNA extraction and had been enrolled into a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis by using state of the art metagenomics technology.
- Colo Rectal Cancer: 29 subjects that exactly meet our inclusion & exclusion criteria were recruited. Demographic and clinical data were entered for each during the introduction to the study and verifying acceptance to participate. Then after unified bowel preparation protocol, a full Colonoscopy was performed after signing the consent, during which mucosal washing samples were collected from the unified 4 colonic segment sites, as specified in methodology.
  Recruitment were completed on 28/05/2012, and all have been identified as sufficient DNA extraction.
  Now, all are identified as sufficient DNA extraction and had been enrolled into a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis by using state of the art metagenomics technology.
- Control: Normal Subjects: 50 subjects that exactly meet our inclusion & exclusion criteria were recruited. Demographic and clinical data were entered for each during the introduction to the study and verifying acceptance to participate. Then after unified bowel preparation protocol, a full Colonoscopy was performed after signing the consent, during which mucosal washing samples were collected from the unified 4 colonic segment sites, as specified in methodology.
  Recruitment were completed on 22/12/2010, however, in view of insufficient DNA extraction of 6 subjects they have been replaced on 19/09/2012 with other 6 subjects following exactly the same protocol.
  Now, all are identified as sufficient DNA extraction and had been enrolled into a comprehensive analysis of the gastrointestinal tract microbiota and its contribution on gut homeostasis by using state of the art metagenomics technology.
Period: Overall Study
Arm/Group | Irritable Bowel Syndrome | Ulcerative Colitis | Crohn's Disease | Colo Rectal Cancer | Control: Normal Subjects
Started | 50 | 50 | 46 | 29 | 50
Completed | 50 (5 subjects were dropped out because of insufficient DNA extraction and accordingly replaced randomly) | 50 (3 subjects were dropped out because of insufficient DNA extraction and accordingly replaced randomly) | 46 (2 subjects were dropped out because of insufficient DNA extraction and accordingly replaced randomly) | 29 | 50 (6 subjects were dropped out because of insufficient DNA extraction and accordingly replaced randomly)
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irritable Bowel Syndrome | Ulcerative Colitis | Crohn's Disease | Colo Rectal Cancer | Control: Normal Subjects | Total
Number analyzed (Participants) | 50 | 50 | 46 | 29 | 50 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 4 | 11 | 0 | 0 | 15
  Between 18 and 65 years | 45 | 45 | 34 | 23 | 41 | 188
  >=65 years | 5 | 1 | 1 | 6 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.93 (14.505) | 34.42 (12.586) | 25.19 (10.672) | 55.03 (10.137) | 53.58 (12.747) | 42.43 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 24 | 14 | 32 | 135
  Male | 19 | 16 | 22 | 15 | 18 | 90
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 50 | 50 | 46 | 29 | 50 | 225

OUTCOME MEASURES:

1. Primary Outcome: Colonic-Mucosa Associated Microbial Species Per Compiled Participants in 5 Different Arms
Description: The entire mucosal microbial community were profiled using high-throughput DNA sequencing and microarray technology. The microarray approach is based on 16S rRNA gene targeted oligonucleotide allowing the rapid detection of thousands of DNA sequences simultaneously and thus constitutes an ideal tool to generate a comprehensive and holistic view of the gut microbial community in all participants of all study arms.
  Then they will be analysed between different colonic segments in each participant, pooled results of participants in each of the 5 arms will be compared to the measurable outcomes of other arms in general.
Time Frame: 1 - 2 weeks
Population: Each participant colonic mucosal microbiota populations pattern were analysed, and then compared to control to look for specific enrichments. If the DNA extract was not enough for sequencing, then the participant sample was excluded, however analysis calculation was based on all enrolled participants. The number analyzed here represent all enrolled
Measure: Number (95% Confidence Interval); unit: microbial species population
Arm/Group | Irritable Bowel Syndrome | Ulcerative Colitis | Crohn's Disease | Colo Rectal Cancer | Control: Normal Subjects
Number analyzed (Participants) | 48 | 48 | 34 | 29 | 49
microbial species population | 40 [4 to 190] | 30 [9 to 190] | 23 [17 to 189] | 23 [20 to 197] | 41 [41 to 41]

ADVERSE EVENTS:
Arm/Group | Irritable Bowel Syndrome | Ulcerative Colitis | Crohn's Disease | Colo Rectal Cancer | Control: Normal Subjects
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/46 | 0/29 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/46 | 0/29 | 0/50

LIMITATIONS AND CAVEATS:
After completing recruitment, the colonic mucosal washing sampling did not result in enough DNA extract and we had to drop some of the participants for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No